CLINICAL TRIAL: NCT00674609
Title: A Double Blind, Randomized, Parallel Group, Placebo Controlled, Comparative Study of the Efficacy, Safety and Tolerability of Cannabis Based Medicine (CBM) Extracts in Patients With Cancer-related Pain.
Brief Title: A Study of Sativex® for Pain Relief in Patients With Advanced Malignancy
Acronym: SPRAY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Mr Richard Potts/ Clinical Operations Director, GW Pharmaceuticals Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GWCA0101
Record Dates: First submitted 2008-04-28; First posted 2008-05-08 (Estimated); Results first posted 2012-08-13 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Palliative Care; Pain; Cancer
Keywords: Palliative Care; Pain; Cancer
MeSH Terms: conditions — Pain; Neoplasms | interventions — nabiximols; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo
- Sativex (Experimental): Active treatment
  Interventions: Drug: Sativex®
- THC Alone (Experimental): Active treatment
  Interventions: Drug: THC Alone

INTERVENTIONS:
Drug: Placebo — Containing colourants and excipients. Subjects received study medication delivered in 100 µl actuations by a pump action oromucosal spray. Maximum permitted dose was eight actuations in any three hour period and 48 actuations in 24 hours.
  Other Names: GW-4000-01
  Arms: Placebo
Drug: Sativex® — Containing D9 tetrahydrocannabinol (THC), 27 mg/ml: cannabidiol (CBD), 25 mg/ml. Subjects received study medication delivered in 100 µl actuations by a pump action oromucosal spray. Maximum permitted dose was eight actuations in any three hour period and 48 actuations (THC 130 mg:CBD 120 mg) in 24 hours.
  Other Names: GW-1000-02
  Arms: Sativex
Drug: THC Alone — Containing THC, 27 mg/ml, as extract of Cannabis sativa L. Subjects received study medication delivered in 100 µl actuations by a pump action oromucosal spray. Maximum permitted dose was eight actuations in any three hour period and 48 actuations (THC 130 mg) in 24 hours.
  Other Names: GW-2000-02; THC
  Arms: THC Alone

SUMMARY:
The purpose of this study is to determine whether Sativex® and GW-2000-02 are effective in the management of subjects with intractable cancer-related pain.

DETAILED DESCRIPTION:
This is a two week (two days baseline and two weeks treatment period), multicentre, double blind, randomised, placebo controlled, parallel group study to evaluate the efficacy of Sativex® and GW-2000-02 in subjects with cancer-related pain. Subjects are screened to determine eligibility and completed a two-day baseline period. Subjects then return to the centre for assessment, randomisation and dose introduction. All subjects are allowed to continue using all their current medications, provided that the dose remains stable throughout the study period. Their progress is reviewed after seven to 10 days and at the end of the study (day 14 to 20), or upon withdrawal. Subjects in this study are given the opportunity to be enrolled in an open label extension study (GWEXT0101).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent.
* Male or female, age 18 years or above.
* Diagnosed with cancer of any type, which is considered to be terminal.
* Diagnosed with cancer-related pain which is not wholly alleviated with their current strong opioid treatment and whose level of pain measured on a NRS is ³four on at least one occasion per day, during the two day run-in period, leading up to visit 1.
* On strong opioid maintenance therapy for at least seven days prior to the screening visit.
* Willing to abstain from any use of cannabis during the study, other than the study medication.
* No cannabinoids use (cannabis, Marinol® or Nabilone) for at least seven days before Visit 1 and willing to abstain from any use of cannabis during the study.
* Clinically acceptable blood results at the screening visit.
* Able (in the investigators opinion) and willing to undertake and comply with all study requirements.
* Willing to allow their own general practitioner, and consultant if appropriate, to be informed of study participation.
* Willing for the Home Office to be notified of his or her participation in the study (applicable to the UK centres only).

Exclusion Criteria:

* Know history of substance misuse.
* Known or suspected to have had an adverse reaction to cannabinoids causing psychosis or other severe psychiatric illness.
* Received any epidural analgesia within 48 hours prior to study entry.
* Either received, within two weeks of study entry, or due to receive chemotherapy or radiotherapy during the study.
* Unable to give informed consent.
* History of any type of schizophrenia, any other psychotic illness, a serious personality disorder, or other significant psychiatric illness other than depression associated with their chronic pain and/or in response to the underlying condition.
* Currently taking levodopa (Sinemet®, Sinemet plus®, Levodopa®, L-dopa®, Madopar®, Benserazide®).
* Had a serious cardiovascular disorder, including angina, uncontrolled hypertension, or an uncontrolled symptomatic cardiac arrhythmia.
* Significant renal or hepatic impairment, who in the opinion of the investigator, were unsuitable for treatment with study medication.
* History of epilepsy.
* Had oral cavity cancers or whose previous treatments had included radiotherapy to the floor of the mouth.
* Female subjects who were pregnant or lactating or of child-bearing potential and were inadequately protected against conception during the study and for three months thereafter.
* Male subjects who were sexually active and who were not using adequate forms of contraception during the study and for three months thereafter.
* Subjects who had participated in a clinical research study in the past four weeks, prior to study entry.
* Planned travel outside the UK during the study (applicable to the UK centres only).
* Subjects who, in the opinion of the investigator, were unsuitable to participate in the study for any other reason, not mentioned in the entry criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2002-02; Primary Completion 2004-02 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy R Johnson, MB ChB, Principal Investigator — Shropshire and Mid-Wales Hospice
Locations (1):
- Shropshire and Mid-Wales Hospice, Shrewsbury, United Kingdom

REFERENCES:
- [Result] Johnson JR, Burnell-Nugent M, Lossignol D, Ganae-Motan ED, Potts R, Fallon MT. Multicenter, double-blind, randomized, placebo-controlled, parallel-group study of the efficacy, safety, and tolerability of THC:CBD extract and THC extract in patients with intractable cancer-related pain. J Pain Symptom Manage. 2010 Feb;39(2):167-79. doi: 10.1016/j.jpainsymman.2009.06.008. Epub 2009 Nov 5. PMID 19896326

RESULTS

PARTICIPANT FLOW:
Groups:
- Sativex: Each 100 uL actuation contained 27 mg/ml THC and 25 mg/ml CBD
- THC Alone: Each 100 uL actuation contained 27 mg/ml THC
- Placebo: Each 100 uL actuation contained colourant and excipients
Period: Overall Study
Arm/Group | Sativex | THC Alone | Placebo
Started | 60 | 58 | 59
Completed | 48 | 45 | 51
Not Completed | 12 | 13 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sativex | THC Alone | Placebo | Total
Number analyzed (Participants) | 60 | 58 | 59 | 177
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 38 | 38 | 115
  >=65 years | 21 | 20 | 21 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (12.08) | 61.3 (12.5) | 60.1 (12.31) | 60.2 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 27 | 82
  Male | 33 | 30 | 32 | 95
Region of Enrollment [Number; unit: participants]
  United Kingdom | 22 | 18 | 21 | 61
  Belgium | 4 | 4 | 3 | 11
  Romania | 34 | 36 | 35 | 105

OUTCOME MEASURES:

1. Primary Outcome: The Change in Mean Pain Numerical Rating Scale (NRS) Score From Baseline to the End of the Treatment.
Description: The pain NRS was complete at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate the number that best describes your pain or average pain in the last 24 hours" where 0 = no pain and 10 = pain as bad as you can imagine. No pain relates to the time prior to the onset of pain due to cancer. A negative value indicates an improvement in pain score from baseline.
Time Frame: 2 weeks: baseline - end of week 2 (last 3 days of treatment)
Population: All subjects who were randomised, received at least one actuation of study medication and had on-treatment efficacy data were included in the ITT population. This population was used for the primary analysis. Presented below is the adjusted mean change from baseline in mean pain NRS.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sativex: Each 100 μl actuation of Sativex delivered a dose containing 2.7 mg THC and 2.5 mg CBD. The maximum permitted dose of study medication was eight actuations in any three hour period, and 48 actuations (130 mg THC and 120 mg CBD) in any 24 hour period.
- THC Alone: Each 100 μl actuation of THC delivered a dose containing 2.7 mg THC only. The maximum permitted dose of study medication was eight actuations in any three hour period, and 48 actuations (130 mg) in any 24 hour period.
- Placebo: Each actuation of placebo delivered the excipients plus colourants. The maximum permitted dose of study medication was eight actuations in any three hour period, and 48 actuations in any 24 hour period.
Arm/Group | Sativex | THC Alone | Placebo
Number analyzed (Participants) | 53 | 52 | 56
units on a scale | -1.32 (1.64) [-1.44 to -0.14] | -0.93 (1.15) [-1.02 to 0.19] | -0.73 (1.51)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change in mean pain NRS score (average pain) was analyzed using analysis of covariance (ANCOVA) with the baseline value as a covariate and region and treatment group as factors. The null hypothesis was that of no treatment difference; Test type: Superiority or Other; p = 0.014, ANCOVA; estimated mean treatment difference = -0.67, 95% CI 2-sided [-1.21 to -0.14]
Statistical Analysis 2: Comparison: THC Alone vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.244, ANCOVA; Estimated mean treatment difference = -0.32, 95% CI 2-sided [-0.86 to 0.22]

2. Secondary Outcome: Sleep Disturbance 0-10 Numerical Rating Scale
Description: The sleep disruption NRS was completed at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate how your pain disrupted your sleep last night?" where 0 = did not disrupt sleep and 10 = completely disrupted (unable to sleep at all). A negative value indicates an improvement in sleep disruption score from baseline.
Time Frame: 2 weeks: baseline to end of week 2 (last 3 days of treatment)
Population: All subjects who were randomised, received at least one actuation of study medication and had on-treatment efficacy data were included in the ITT population, used for this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | THC Alone | Placebo
Number analyzed (Participants) | 54 | 54 | 56
units on a scale | -0.59 (1.88) [-0.97 to 0.34] | -0.25 (2.33) [-0.64 to 0.68] | -0.21 (1.72)
Statistical Analysis 1: Comparison: Sativex vs Placebo; Each secondary variable was tested using a two-sided significance level of α=0.05, unless otherwise specified. P-values of < 0.05 were considered statistically significant. If the overall treatment effect for the secondary variables was statistically significant then treatment comparisons was made between active treatments and placebo; Test type: Superiority or Other; p = 0.346, ANCOVA; Estimated mean treatment difference = -0.31, 95% CI 2-sided [-0.97 to 0.34]
Statistical Analysis 2: Comparison: THC Alone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.95, ANCOVA; Estimated mean treatment difference = 0.02, 95% CI 2-sided [-0.64 to 0.68]

3. Secondary Outcome: Nausea 0-10 Numerical Rating Scale
Description: The nausea NRS was completed at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate how sick you felt throughout the day?" where 0 = not sick at all and 10 = very sick. A negative value indicates an improvement in nausea score from baseline.
Time Frame: 2 weeks; baseline - end of week 2 (last 3 days of treatment)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | THC Alone | Placebo
Number analyzed (Participants) | 54 | 54 | 56
units on a scale | 0 (2.19) [-0.11 to 1.09] | 0.27 (1.83) [-0.13 to 1.05] | -0.16 (1.25)
Statistical Analysis 1: Comparison: Sativex vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.11, ANCOVA; Estimated mean treatment difference = 0.49, 95% CI 2-sided [-0.11 to 1.09]
Statistical Analysis 2: Comparison: THC Alone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.126, ANCOVA; Estimated mean treatment difference = 0.46, 95% CI 2-sided [-0.13 to 1.05]

4. Secondary Outcome: Memory 0-10 Numerical Rating Scale
Description: The memory NRS was completed at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate how well you are able to remember what you have done in the past 24 hours?" where 0 = very well and 10 = not at all. A negative value indicates an improvement in memory score from baseline.
Time Frame: 2 weeks: baseline - end of week 2 (last 3 days of treatment)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | THC Alone | Placebo
Number analyzed (Participants) | 54 | 54 | 56
units on a scale | 0.58 (2.06) | 0.57 (1.90) | 0 (1.35)
Statistical Analysis 1: Comparison: Sativex vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.045, ANCOVA; Estimated mean treatment difference = 0.65, 95% CI 2-sided [0.01 to 1.28]
Statistical Analysis 2: Comparison: THC Alone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.053, ANCOVA; Estimated mean treatment difference = 0.62, 95% CI 2-sided [-0.01 to 1.25]

5. Secondary Outcome: Appetite 0-10 Numerical Rating Scale
Description: The appetite NRS was completed at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate how your appetite has been throughout the day?" where 0 = very good and 10 = very poor. A negative value indicates an improvement in appetite score from baseline.
Time Frame: 2 weeks: baseline - end of week 2 (last 3 days of treatment)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | THC Alone | Placebo
Number analyzed (Participants) | 54 | 54 | 56
units on a scale | 0.24 (2.29) | 0.18 (1.91) | -1.65 (1.94)
Statistical Analysis 1: Comparison: Sativex vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.016, ANCOVA; estimated mean treatment difference = 0.83, 95% CI 2-sided [0.16 to 1.51]
Statistical Analysis 2: Comparison: THC Alone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.056, ANCOVA; Estimated mean treatment difference = 0.66, 95% CI 2-sided [-0.02 to 1.33]

6. Secondary Outcome: Concentration 0-10 Numerical Rating Scale
Description: The concentration NRS was completed at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate how well have you been able to concentrate throughout the day e.g. when reading a newspaper?" where 0 = very well and 10 = not at all. A negative value indicates an improvement in concentration score from baseline.
Time Frame: 2 weeks: baseline - end of week 2 (last 3 days of treatment)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | THC Alone | Placebo
Number analyzed (Participants) | 54 | 54 | 56
units on a scale | 0.26 (1.66) | 0.22 (1.80) | -0.32 (1.39)
Statistical Analysis 1: Comparison: Sativex vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.021, ANCOVA; Estimated mean treatment difference = 0.68, 95% CI 2-sided [0.10 to 1.25]
Statistical Analysis 2: Comparison: THC Alone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.028, ANCOVA; Estimated treatment difference = 0.64, 95% CI 2-sided [0.07 to 1.22]

7. Secondary Outcome: EORTC Quality of Life Questionnaire (EORTC-QLQC30)
Description: Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30), a core cancer-specific questionnaire containing 30 items on patients' functioning, global quality of life, disease- and treatment related symptoms. Higher scores indicate a greater degree of symptoms, min.: 0, Max.: 100
Time Frame: 2 weeks; baseline and end of treatment (2 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | THC Alone | Placebo
Number analyzed (Participants) | 49 | 50 | 52
units on a scale | 4.93 (17.51) | 3.57 (18.32) | 4.74 (18.50)
Statistical Analysis 1: Comparison: Sativex vs Placebo; Analysis of the change from baseline was assessed using ANCOVA, adjusting for the effects of the baseline value. The significance of the treatment effect, after adjusting for the baseline value, was assessed using the F-test from the ANCOVA. If found significant at the 5% level, then the mean difference between treatments together with 95% CI were presented; Test type: Superiority or Other; p = 0.443, ANCOVA; estimated mean treatment difference = 2.47, 95% CI 2-sided [-3.87 to 8.81]
Statistical Analysis 2: Comparison: THC Alone vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.793, ANCOVA; estimated mean treatment difference = 0.84, 95% CI 2-sided [-5.46 to 7.13]

8. Secondary Outcome: Brief Pain Inventory Short Form
Description: The BPI-SF is a 14-item questionnaire that asks patients to rate pain over the prior week and the degree to which it interferes with activities on a 0 to 10 scale, where 0=no pain and 10=pain as bad as you can imagine. Severity is measured as worst pain, least pain, average pain, and pain right now. The severity composite score was calculated as the arithmetic mean of the four severity items(range 0-10). The minimum value is zero and maximum is 10. A higher score represents a poor outcome.
Time Frame: End of 2 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | THC Alone | Placebo
Number analyzed (Participants) | 15 | 17 | 18
units on a scale | 0.2 (5.63) | -3.38 (6.43) | 0.41 (5.55)
Statistical Analysis 1: Comparison: Sativex vs Placebo; Change in pain scores on-treatment were be compared between groups using analysis of covariance (ANCOVA). The baseline pain score was fitted as a covariate in the model. The significance of the treatment effect after adjusting for baseline pain score was assessed using the F-test from the ANCOVA. If this was significant at the 5% level, then the mean difference between treatments together with the 95% confidence interval was presented for Sativex versus placebo and THC versus placebo; Test type: Superiority or Other; p = 0.619, ANCOVA; Estimated mean treatment difference = -1.04, 95% CI 2-sided [-5.23 to 3.15]
Statistical Analysis 2: Comparison: THC Alone vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.048, ANCOVA; Estimated mean treatment difference = -4.07, 95% CI 2-sided [-8.10 to -0.05]

9. Primary Outcome: The Consumption of Escape Analgesic Medication.
Description: Subjects recorded their use of escape medication each day on their diary card.
Time Frame: 2 weeks: baseline - end of week 2 (last 3 days of treatment)
Population: The primary population for this analysis was the intention-to-treat (ITT) population, which included all randomised subjects who received at least 1 dose of study medication and had on-treatment efficacy data. The primary analysis escape medication usage i.e. the number of days escape medication was used did not include any covariates.
Measure: Mean (Standard Deviation); unit: tablets per day
Arm/Group | Sativex | THC Alone | Placebo
Number analyzed (Participants) | 54 | 52 | 57
tablets per day | 0.72 (0.821) [-0.25 to 0.16] | 0.88 (0.852) [-0.19 to 0.22] | 0.68 (0.662)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The on-treatment data was calculated from all available data during the last three days. The number of days the escape medication was used out of the last three days taken in the study was compared between treatments using logistic regression with a cumulative logit model. From this analysis the frequency distribution (%) of number days escape medication was used was presented together with the odds ratio, p-value and 95% CI for the treatment contrasts; Test type: Superiority or Other; p = 0.688, Regression, Logistic; estimated mean treatment difference = -0.04, 95% CI 2-sided [-0.25 to 0.16]
Statistical Analysis 2: Comparison: THC Alone vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.899, Regression, Logistic; Estimated mean treatment difference = 0.01, 95% CI 2-sided [-0.19 to 0.22]

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring from the time of consent to post study follow up (14 - 20 days) were collected. All deaths and serious adverse events (SAEs) occurring within 28 days of the final dose of study medication were also collected.
Description: All AEs occurring during the study were reported on the running logs at the back of the study case report form.
Groups:
- Sativex: Maximum number of daily sprays was 48 giving a maximum daily dose of 130 mg THC and 120 mg CBD
- THC Alone: Maximum number of daily sprays was 48 giving a maximum daily dose of 130 mg THC
- Placebo: Maximum number of daily sprays was 48
Arm/Group | Sativex | THC Alone | Placebo
Serious Adverse Events (participants affected / at risk) | 13/60 | 13/58 | 7/59
Other Adverse Events (participants affected / at risk) | 51/60 | 45/58 | 44/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sativex (N=60) | THC Alone (N=58) | Placebo (N=59)
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 | 0 (0)
Nausea aggravated (Gastrointestinal disorders) | 1 | 0 (0) | 0 (0)
Disease progression nos (General disorders) | 1 | 1 | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1
Malaise (General disorders) | 0 (0) | 1 | 0 (0)
Weakness (General disorders) | 1 | 0 (0) | 0 (0)
Bronchopneumonia nos (Infections and infestations) | 0 (0) | 1 | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 | 0 (0)
Blood urine present (Investigations) | 1 | 0 (0) | 0 (0)
Hyperglycaemia nos (Metabolism and nutrition disorders) | 0 (0) | 1 | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1
Neoplasm progression nos (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2
Metastases to brain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 | 0 (0)
Metastases to prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 | 0 (0)
Spinal cord compression nos (Nervous system disorders) | 1 | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 2 | 1
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1
Disorientation (Psychiatric disorders) | 0 (0) | 1 | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 | 0 (0) | 0 (0)
Renal Failure nos (Renal and urinary disorders) | 0 (0) | 1 | 0 (0)
Dyspnoea nos (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1
Family stress nos (Social circumstances) | 0 (0) | 0 (0) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=60) | THC Alone (N=58) | Placebo (N=59)
Somnolence (Nervous system disorders) | 9 | 8 | 8
Nausea (Gastrointestinal disorders) | 7 | 6 | 6
Dizziness (Nervous system disorders) | 7 | 7 | 3
Neoplasm progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5 | 3
Vomiting (Gastrointestinal disorders) | 5 | 4 | 4
Confusion (Psychiatric disorders) | 4 | 0 | 2
Diarrhoea NOS (Gastrointestinal disorders) | 4 | 0 | 2
Constipation (Gastrointestinal disorders) | 3 | 0 | 6
Liver function test NOS abnormal (Investigations) | 3 | 0 | 2
Weakness (General disorders) | 3 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 0 | 1
Hypotension NOS (Vascular disorders) | 3 | 0 | 0
Urinary retention (Renal and urinary disorders) | 3 | 0 | 0
Oral pain (General disorders) | 0 | 5 | 3
Glossodynia (General disorders) | 0 | 5 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 5 | 3
Fatigue (General disorders) | 0 | 3 | 0
Chest Pain (General disorders) | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications, for example manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.